CLINICAL TRIAL: NCT02987595
Title: Effects of Lignan-rich Diet on Cardiometabolic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Responsible Party: Principal Investigator, Dr. Rikard Landberg, Associate professor, Head of Unit Food and Health, Department of Food Science, Swedish University of Agricultural Sciences (SLU), Swedish University of Agricultural Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SwedishUAS
Record Dates: First submitted 2015-06-16; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Syndrome; Overweight; Central Obesity; Impaired Glucose Tolerance
Keywords: intervention; lignans; whole-grain
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity, Abdominal; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole-grain rye then wheat (Experimental): Whole-grain rye, high lignan Whole-grain rye products for 8 weeks, then a wash-out period of 8 weeks, and then whole-grain wheat products for 8 weeks
  Interventions: Other: Whole-grain rye, high lignan; Other: Whole-grain wheat, low lignan
- Whole-grain wheat then rye (Experimental): Whole-grain wheat, low lignan Whole-grain wheat products for 8 weeks, then a wash-out period of 8 weeks, and then whole-grain rye products for 8 weeks
  Interventions: Other: Whole-grain rye, high lignan; Other: Whole-grain wheat, low lignan

INTERVENTIONS:
Other: Whole-grain rye, high lignan — Intervention week 1-8: 50 g rolled rye + 50 g puffs + 4 pieces of crisp bread + 70 g pasta. Additionally for intervention week 4-8: 4 lignan capsules per day
Other: Whole-grain wheat, low lignan — Intervention week 1-8: 100 g puffs + 4 pieces of crisp bread + 70 g pasta.

SUMMARY:
Diet plays an important role in relation to prevention of type 2 diabetes, cardiovascular disease and certain cancers. Studies have shown that diets with high whole-grain content could decrease the risk of these lifestyle related diseases and in Sweden the national dietary guidelines recommends whole-grain based instead of refined cereal products. It is, however, not clear whether whole-grain from wheat and rye share similar protective effects since there are large differences in amount and quality of dietary fibre and associated bioactive compounds. The aim of this study is to evaluate the impact of a wholegrain diet with low- or high lignan content on different cardiometabolic risk factors with the primary endpoint being blood glucose levels after 2h oral glucose tolerance test in men with metabolic syndrome or sign thereof.

DETAILED DESCRIPTION:
The study will be conducted in a randomized, cross-over design (8 wk intervention periods). The lignan-rich diet will be based on whole-grain rye products whereas the control diet will be based on whole-grain wheat products with some added wheat bran. Both diets will provide similar amount of whole grain (g/d) and total dietary fiber content (but dietary fibre quality will be different). Although rye has high lignan content, the aim is to further increase the lignan intake half-way through the whole grain rye intervention period. This will allow us to distinguish the effect of lignans from the effect of whole grain rye as well as evaluating potential differences in effects on cardiometabolic risk factors between whole grain wheat and whole grain rye intake after 4-week consumption. The study design will also allow us to investigate the effects of a putative interaction between microbiome x lignan rich diet and its implication of metabolic risk factors.

Blood samples will be collected by trained nurses at screening, baseline, after 4 weeks and 8 weeks of first intervention period, after wash-out (8 weeks), and after 4 weeks and 8 weeks of the second intervention period.

At each examination day participants will arrive to the test laboratory for blood samples and an oral glucose tolerance test (OGTT) where participants will be given a drink with 75 g of glucose to consume within 10 minutes. Blood samples will be taken after 30, 60 and 120 minutes. Furthermore, participants will be instructed to complete one 3-day weighted food record and also to collect 24-h urine and a fecal sample at week 0, 4, 8, 16, 20 and 24.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 kg/m2
* waist circumference > 102 cm
* at least one of the following: blood pressure >130/85 mmHg, serum triglycerides ≥1.69 mmol/L; HDL cholesterol <1.04 mmol/L; or serum glucose ≥6.1 mmol/L

Exclusion Criteria:

* smokers
* antibiotic use past 6 months
* cancer diagnose (past 5 years) or other chronic disease diagnosis
* excessive alcohol consumption (>21 units/week)

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels | 8 weeks

SECONDARY OUTCOMES:
Blood lipids | 8 weeks
Inflammatory markers | 8 weeks
Oxidative stress markers | 8 weeks
Enterolignans in blood and urine | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Principal Investigator — Swedish University of Agricultural Sciences
Locations (1):
- Paediatric Research Facility; The Children's Hospital at Uppsala University Hospital, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Eriksen AK, Brunius C, Mazidi M, Hellstrom PM, Riserus U, Iversen KN, Fristedt R, Sun L, Huang Y, Norskov NP, Knudsen KEB, Kyro C, Olsen A, Tjonneland A, Dicksved J, Landberg R. Effects of whole-grain wheat, rye, and lignan supplementation on cardiometabolic risk factors in men with metabolic syndrome: a randomized crossover trial. Am J Clin Nutr. 2020 Apr 1;111(4):864-876. doi: 10.1093/ajcn/nqaa026. PMID 32097450